CLINICAL TRIAL: NCT01052610
Title: Assessment of Effectiveness and Safety of Annual Sublingual Immunotherapy in Children With Bronchial Asthma and/or Allergic Rhinitis Allergic to House Dust Mites
Brief Title: Assessment of Sublingual Immunotherapy in Children Allergic to House Dust Mites
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Iwona Stelmach, MD, PhD, Professor, Medical University of Lodz
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 502-12-760, 503-2056-1
Record Dates: First submitted 2010-01-12; First posted 2010-01-20 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Bronchial Asthma; Allergic Rhinitis
Keywords: SLIT; bronchial asthma; allergic rhinitis
MeSH Terms: conditions — Asthma; Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active group (Active Comparator): Group of children with bronchial asthma and/ or allergic rhinitis 6-18 years old receiving annually house dust mites sublingual allergen extract
  Interventions: Drug: sublingual house dust mites allergen extract
- Placebo group (Placebo Comparator): Group of children with bronchial asthma and/or allergic rhinitis 6-18 years old receiving placebo in sublingual applicator
  Interventions: Drug: placebo in sublingual applicator

INTERVENTIONS:
Drug: sublingual house dust mites allergen extract — Staloral 300 IR, Stallergenes, France
  Arms: Active group
Drug: placebo in sublingual applicator — placebo for Staloral 300 IR, Stallergenes, France
  Arms: Placebo group

SUMMARY:
The purpose of the trial is to asses the efficacy and safety of sublingual annual immunotherapy in children with bronchial asthma and/or allergic rhinitis allergic to house dust mites.

DETAILED DESCRIPTION:
Allergen immunotherapy is currently the only one method of cause treatment of the IgE-dependent allergic diseases. Sublingual immunotherapy (SLIT) is the method which allows to give allergens via alternative oral route in patients home. Due to possibility of avoiding injection this therapy offers better relationship with pediatric patient. However efficacy and safety of sublingual immunotherapy are still important issues, especially in asthmatic children. The purpose of the trial is to asses the efficacy and safety of sublingual annual immunotherapy in children with bronchial asthma and/or allergic rhinitis allergic to house dust mites.

ELIGIBILITY:
Inclusion Criteria:

* patients with bronchial asthma and/or allergic rhinitis allergic to house dust mites first diagnosed at least 2 years before the study

Exclusion Criteria:

* active respiratory tract infection requiring antibiotic treatment within 4 weeks before the study
* hospitalisation due to asthma exacerbation during the 3 months before the first visit
* known contraindications of SIT according to the EAACI
* previous allergen immunotherapy
* use of systemic corticosteroids
* other clinically significant pulmonary, hematologic, hepatic, gastrointestinal, renal, endocrine, neurologic, cardiovascular, and/or mental diseases or malignancy that either put the patient at risk when participating in the study or could influence the results of the study

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms of asthma and allergic rhinitis and use of rescue medication | Visit No 2 (before SLIT),VISIT No 4(after 1 year of SLIT), Visit No 6(after 3 years of SLIT)

SECONDARY OUTCOMES:
Change of percent of regulatory lymphocytes in peripheral blood | Visit No 2 (before SLIT),VISIT No 4(after 1 year of SLIT), Visit No 6(after 3 years of SLIT)
assessment of inflammatory markers in exhaled breath condensate and FeNO | Visit No 2 (before SLIT),VISIT No 4(after 1 year of SLIT), Visit No 6(after 3 years of SLIT)
non-specific bronchial hyperreactivity with methacholine (PC20M), specific conjunctival provocation test | Visit No 2 (before SLIT),VISIT No 4(after 1 year of SLIT), Visit No 6(after 3 years of SLIT)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona Stelmach, MD, PhD, Prof, Study Chair — Department of Pediatrics and Allergy
Locations (1):
- Department of Pediatrics and Allergy, Lodz, Poland